CLINICAL TRIAL: NCT05777447
Title: Long Term Results of Aorto-iliac Mycotic Aneurysms
Brief Title: International Multicenter Mycotic Aneurysm Aorto-iliac Study
Acronym: MAAI
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, TINELLI GIOVANNI, Prof, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2855
Record Dates: First submitted 2023-03-09; First posted 2023-03-21 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Mycotic Aneurysm; Aortic Diseases
MeSH Terms: conditions — Aneurysm, Infected; Aortic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Mycotic aortic-iliac aneurysms and in situ reconstruction — Surgical treatment of mycotic aortic-iliac aneurysms and in situ reconstruction

SUMMARY:
The term mycotic aneurysm (MA) is commonly used to describe all infected aneurysms. Although MAs are believed to occur uncommonly, the true incidence is difficult to determine and is probably underestimated since MAs can be asymptomatic and are diagnosed only at autopsy. In an autoptic study, mycotic aortic aneurysms (MAAs) were reported in 3.3% of all detected aneurysms. The incidence of infected aneurysms of the aorta and iliac arteries ranges from 0.6% to 1.3%.

A recent literature review of the management of MAAs showed that therapeutic strategies are multiple, including open surgical repair (OSR) in the majority of cases, endovascular aortic repair (EVAR), which increased over the last decade, and medical treatment alone for patients unfit for any aortic repair in a very limited part. Following the unfavorable prognosis towards rupture and since the medical treatment alone in mycotic aneurysms has shown mortality of almost 100%, surgical treatment is generally the preferred option.

Surgical treatment includes both open and endovascular surgery. The latter is less invasive than conventional surgery but does not involve resection of the infected tissue and is therefore associated with an increased risk of sepsis and prosthesis infection. The gold standard is still open surgery, including extra-anatomic reconstruction and in situ repair, with different type of vascular graft.

This is a multicenter retrospective observational study. It will examine all patients undergoing surgical treatment of mycotic aortic-iliac aneurysms and in situ reconstruction at the participating centers.

ELIGIBILITY:
Inclusion Criteria:

* primary mycotic aorto-iliac aneurysm who underwent in situ repair

Exclusion Criteria:

* patient with vascular graft infections;
* patient with secondary aorto-enteric fistula.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing surgical treatment of mycotic aortic-iliac aneurysms and in situ reconstruction at the participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Early mortality | Mortality within 30 days after surgery
  Mortality after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No